CLINICAL TRIAL: NCT04703569
Title: Effect of Compressive Therapies on the Healing of Venous Ulcers in Primary Health Services: Randomized Clinical Trial
Brief Title: Effect of Compressive Therapies on the Healing of Venous Ulcers
Acronym: VENOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Casex Innovation in Healthcare (Unknown); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16087119.2.0000.5327
Record Dates: First submitted 2020-12-17; First posted 2021-01-11 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Venous Ulcers
Keywords: Varicose Ulcer; Compression Bandages; Wound Healing; Nursing; Primary Health Care; Intervention study; Cost-effectiveness
MeSH Terms: conditions — Varicose Ulcer | interventions — Bandages

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monolayer high compression elastic bandage (Experimental): An elastic bandage of cotton, viscose, nylon and elastane
  Interventions: Procedure: Dressing with monolayer high compression elastic bandage
- Unna boot (Active Comparator): A wet bandage with zinc oxide
  Interventions: Procedure: Dressing with Unna boot

INTERVENTIONS:
Procedure: Dressing with monolayer high compression elastic bandage — The nurse will be apply the therapy high compression elastic bandage once a week, during 26 weeks
  Arms: Monolayer high compression elastic bandage
Procedure: Dressing with Unna boot — The nurse will be apply the therapy Unna Boot once a week, during 26 weeks.
  Arms: Unna boot

SUMMARY:
The objective of the study is to compare the effect of two treatments on the healing of venous ulcers in follow-up people in two Primary Health Services, in a city in southern Brazil. The two treatments that will be tested are: (1) the high compression elastic bandage and (2) Unna boot. The two treatments are indicated for the treatment of people with venous insufficiency and who have an active ulcer. The treatment will last 26 weeks (6 months). Once a week, during 26 weeks, a nurse will perform the dressing and will apply the therapy high compression elastic bandage or Unna boot according to a drawing and in every two weeks an evaluator will assess the characteristics of the ulcers and the size.

DETAILED DESCRIPTION:
The primary objective is to compare the effect of two compressive therapies, high compression elastic bandage and Unna boot, on time and on the healing characteristics of venous ulcers in Primary Health Care and the secondary objectives are to verify the effects of the therapies in tissue integrity and at the level of pain, to identify quality of life of the participants and to evaluate the cost-effectiveness of the two therapies from the perspective of the Unified Health System. A randomized clinical trial is being carried out in two Primary Health Services in Porto Alegre city, with people with active venous ulcer. 126 venous ulcers, 63 in each group will be followed. The A group receives elastic compressive therapy (high compression elastic bandage) and the B group receives inelastic compressive therapy (Unna boot) by randomization. Once a week, during 26 weeks, a nurse applies the therapy according to the randomization group. And a blind evaluator for therapies will assess the characteristics of the ulcers and the size, on the first day and in every two weeks until 26ª week.

ELIGIBILITY:
Inclusion Criteria:

* people with diagnosis of chronic venous insufficiency recorded in medical records, with active venous ulcer;
* with indication of compressive therapy, who are not using any of the therapies used in the study and who have not used them within 30 days of the initial moment of data collection;
* 18 years old or older;
* with Ankle-Brachial Index (ABI) between 0.8 and 1.2;
* with pulses present on palpation in lower limbs;
* walking people;
* with Body Mass Index (BMI) between ≥ 18.5 kg/m2 and 39.9 kg/m2 (for elderly people: ≥ 22 kg/m2 and 39.9 kg/m2);
* with ankle circumference greater than 18cm.

Exclusion Criteria:

* pregnant women;
* people with mixed, infected or in the epithelialization phase UV (with epithelial tissue in 90% of the UV area);
* uncontrolled diabetics (with Glycated Hemoglobin greater than 7% in the last six months);
* people with medical diagnosis of dermatological, rheumatological and oncological diseases in the member of the active UV or immunosuppressive diseases (for influencing the healing process);
* with allergy to any f the components of the compressive therapies used in the study;
* people using immunosuppressants and/or corticosteroids for more than 21 days (for influencing the healing process).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Effect of the therapies on time and on the healing characteristics of venous ulcers | On first day and in every two weeks, during 26 weeks.
  A blind evaluator for therapies will assess the characteristics of the ulcers using a Likert scale, being 1 the worst score and 5 best score, proposed to Nursing Outcomes Classification (NOC), in the outcome Wound Healing: Secondary Intention. This outcome has indicators to assess the healing characteristics, such as granulation tissue; necrosis; epithelial tissue; exsudate; erythema; oedema; macerated skin; odor and planimetry.

SECONDARY OUTCOMES:
The effects of the therapies at the level of pain | On first day and in every two weeks, during 26 weeks.
  A blind evaluator for therapies will ask about of the pain on the first day and in every two weeks.
Cost-effectiveness of the therapies | 26 weeks
  Direct costs to perform the dressing will be measured through a tool built by the researches. Every week, the nurses will take notes of all products they used and the time spent to perform the dressing (using a stopwatch). This will be converted into monetary value. Besides that, a blind evaluator for therapies will assess the effectiveness through the wound planimetry. In the end, the relationship between cost-effectiveness will be calculated.
Health-related quality of life | On first day, on the 12ª week and on the 26ª week.
  The SF-6D Questionnaire will be applied to the participants to identify the quality of life, on the first day, on the 12ª week and on the 26ª week. The Short Form-6 Dimension (SF-6D) is a widely used preference-based generic health-related quality of life measure with a multiattribute classification system consisting of six dimensions: physical functioning, role functioning, social functioning, pain, mental health, and vitality. Each dimension is composed of three to five levels. The SF-6D values range from 0.315 to 1, with higher scores indicating better health-related quality of life anchoring on the 0 (dead) to 1 (full health) scale.
The effects of the therapies at the tissue integrity | On first day and in every two weeks, during 26 weeks.
  A blind evaluator for therapies will assess the tissue integrity using a Likert scale, being 1 the worst score and 5 best score, proposed to Nursing Outcomes Classification (NOC), in the outcome Tissue Integrity: Skin and Mucous Membranes. This outcome has indicators to assess the tissue integrity, such as necrosis; skin hydration and skin pigmentation.

CONTACTS AND LOCATIONS:
Overall Officials: Lisiane Paskulin, PhD, Study Director — Federal University of Rio Grande do Sul
Locations (3):
- Brazil (3):
  - Unidade de Saúde Modelo, Porto Alegre, Rio Grande do Sul
  - Unidade de Saúde Santa Cecília, Porto Alegre, Rio Grande do Sul
  - Unidade de Saúde Santa Marta, Porto Alegre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cordova FP, Fuhrmann AC, Machado, DO, Mocellin D, Silva BU, Lucena AF, Paskulin LMG. Clinical and economic analysis on compression treatment of venous leg ulcers: clinical trial protocol VENOS. Wound Practice and Research. 2022; 30(4): 216-222.
- See also: Article — https://journals.cambridgemedia.com.au/wpr/volume-30-number-4/clinical-and-economic-analysis-compression-treatment-venous-leg-ulcers-clinical-trial-protocol-venos